CLINICAL TRIAL: NCT07365930
Title: Non-Interventional Study on the Benefits of Transjugular Intrahepatic Portosystemic Shunting in Patients With Hepatocellular Carcinoma Receiving Atezolizumab Plus Bevacizumab in First-Line Therapy
Brief Title: NIS on the Benefits of TIPS in Patients With HCC Receiving Atezo+Bev in 1st-Line Therapy
Acronym: NISTIPS
Status: Recruiting | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Roche Pharma AG (Industry); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: NISTIPS TRITICC-4; ML46195 (Other: Roche)
Record Dates: First submitted 2025-12-09; First posted 2026-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; TIPS; Tecentriq; Avastin; transjugular intrahepatic portosystemic shunting; Hepatocellular carcinoma; observational study; non-interventional study; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC patients in atezo+bev treatment without TIPS: Out of 350 HCC patients 168 patients with histologically confirmed, locally advanced or metastatic and/or unresectable liver cancer, without prior transjugular intrahepatic portosystemic shunting and receiving atezolizumab + bevacizumab treatment, will be assigned to analysis cohort 1: HCC patients in atezo+bev treatment without TIPS
- HCC patients in atezo+bev treatment with TIPS: Out of 350 HCC patients 182 patients with histologically confirmed, locally advanced or metastatic and/or unresectable liver cancer, with prior transjugular intrahepatic portosystemic shunting and receiving atezolizumab + bevacizumab treatment, will be assigned to analysis cohort 1: HCC patients in atezo+bev treatment with TIPS

SUMMARY:
The NISTIPS TRITICC-4 study is a prospective, multicentre, non-interventional cohort study to analyze the effectiveness of transjugular intrahepatic portosystemic shunting (TIPS) in patients with Hepatocellular carcinoma (HCC) receiving atezolizumab plus bevacizumab as first-line treatment. It will further characterize the effectiveness of atezolizumab and bevacizumab therapy, investigate post-market safety and evaluate health-related quality in HCC patient cohorts with or without TIPS in a real-world setting.

DETAILED DESCRIPTION:
While TIPS effectively treats CSPH in cirrhosis, its role in HCC patients receiving systemic therapy remains unclear. The NISTIPS TRITICC-4 study will investigate whether TIPS in patients receiving atezo+bev reduces portal hypertension-related complications and improves therapy outcomes. We hypothesize that TIPS is feasible in non-resectable HCC, lowers the risk of hepatic decompensation, and improves survival and treatment effectiveness by preserving liver function. Furthermore, an observational cohort study like NISTIPS TRITICC-4 offers an opportunity to evaluate the effectiveness, safety and tolerability of atezo+bev treatment with or without TIPS in a more heterogeneous patient population, by capturing data on treatment outcomes, quality of life, and safety in daily clinical practice. Moreover, it helps to identify patient subgroups, which may derive benefits or experience specific risks, helping to optimize personalized treatment strategies.

The NISTIPS TRITICC-4 study is a prospective, multicentre, cohort study with associated accompanying research including archival tissue sample collection, which enrolls 350 patients in Germany of both sexes and ages over 18 years. Eligible patients are diagnosed with locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC) in 1st line therapy setting without (Analysis Cohort 1) or with (Analysis Cohort 2) TIPS receiving atezolizumab + bevacizumab according to the market authorization.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a histologically confirmed, locally advanced or metastatic and/or unresectable HCC with:

   1. the presence of liver cirrhosis (cirrhosis confirmed by histology or liver stiffness or with unequivocal signs in ultrasound, endoscopy, and/or blood tests),
   2. a disease that is not amenable to curative surgical and/or locoregional therapies, or a progressive disease after surgical and /or locoregional therapies,
2. A decision for treatment with atezolizumab + bevacizumab according to the market authorization with or without TIPS has been made before enrolling into the study by the treating physician.

NOTE: Patients who have already received 1-2 cycles of atezo+bev therapy are eligible for enrollment into the NISTIPS TRITICC-4 study, when the prescription of the medicine or other therapeutic strategies are clearly separated from the decision to include the patient in the study.

Exclusion Criteria:

1. The patient has not provided signed informed consent.
2. The patient is under 18 years of age at the time of giving signed informed consent.
3. The patient is unable to understand all implications of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NISTIPS TRITICC-4 study enrolls participants in Germany of both sexes and ages over 18 years. Eligible patients are diagnosed with locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC) in 1st line therapy setting without (Analysis Cohort 1) or with (Analysis Cohort 2) TIPS.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2031-12-17 (Estimated); Study Completion 2031-12-17 (Estimated)

PRIMARY OUTCOMES:
Time to deterioration of liver function (TTDL) | up to 72 months
  Time to deterioration of liver function (TTDL) is used as outcome measure to analyze the effectiveness of transjugular intrahepatic portosystemic shunting (TIPS) in patients with Hepatocellular carcinoma (HCC) receiving atezolizumab plus bevacizumab as first-line treatment in a real-world scenario.
  Liver function deterioration is registered if any of the following criteria was met for more than 4 weeks (>28 days in a row):
  * Total bilirubin > 2.0 x ULN OR > 2.0 x baseline if baseline was abnormal
  * Alanine aminotransferase (ALT) AND aspartate aminotransferase (AST) > 5x ULN OR > 5.0 x baseline if baseline was abnormal
  * Alkaline phosphatase >2.5x ULN OR > 2.5 x baseline (if baseline was abnormal)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 72 months
  Overall survival (OS) is used as measurement to further characterize the effectiveness of atezolizumab and bevacizumab therapy in real-world HCC patient cohorts with or without TIPS.
Time on treatment (ToT) | up to 72 months
  Time on treatment (ToT), defined as duration from the first day of atezo+bev therapy to the day of the last dose of atezo+bev therapy
Prevalence of bleeding adverse events | up to 72 months
  Prevalence of bleeding adverse events post-administration of atezo+bev treatment
Overall Response Rate (ORR) | up to 72 months
  Overall Response Rate (ORR) defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), as assessed by the investigator according to local protocol.
Time to New Extrahepatic Lesions or death due to any cause (TTNEL) | up to 72 months
  Time to New Extrahepatic Lesions or death due to any cause (TTNEL) after initiation of atezo+bev treatment
Post-market safety of atezolizumab plus bevacizumab | up to 72 months
  To investigate post-market safety of the authorized treatment with atezolizumab plus bevacizumab in HCC patient cohorts with or without TIPS, type, frequency, causality and severity of adverse events with severity according to NCI CTCAE v5.0 including the rate of TIPS-related complications will be analyzed.
Proportion of patients with improved, maintained, or worsened Health-Related Quality of Life (HR-QoL) according to EORTC QLQ-C30 and QLQ-HCC18 assessment | up to 72 months
  Proportion of patients with improved, maintained, or worsened Health-Related Quality of Life (HR-QoL) scores with a ≥ 10-point change considered clinically meaningful in HR-QoL scores derived from EORTC QLQ-C30 and QLQ-HCC18 assessment is the used measurement to evaluate health-related quality of life in real-world HCC patient cohorts receiving atezolizumab plus bevacizumab as first-line treatment with or without TIPS.
Time to HR-QoL Deterioration (HR-QoL TTD) derived from EORTC QLQ-C30 and QLQ-HCC18 assessment | up to 72 months
  Time to HR-QoL Deterioration (HR-QoL TTD), measured from study enrolment to the first ≥10 points decrease of HR-QoL score compared to baseline HR-QoL score with HR-QoL scores derived from EORTC QLQ-C30 and QLQ-HCC18 assessment, is the used measurement to evaluate health-related quality of life in real-world HCC patient cohorts receiving atezolizumab plus bevacizumab as first-line treatment with or without TIPS.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Roderburg, Professor, Principal Investigator — Heinrich Heine University of Duesseldorf, University Hospital of Duesseldorf
Locations (1):
- University Hospital of Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.